CLINICAL TRIAL: NCT00130689
Title: A Phase II Trial of Cetuximab in Unresectable or Metastatic Esophageal and Gastric Carcinoma
Brief Title: Use of Cetuximab for Unresectable or Metastatic Esophageal and Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Chan, MD, MPH, Overall PI, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-113
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Esophageal Cancer; Gastric Cancer; Neoplasm Metastasis
Keywords: Esophageal Cancer; Gastric Cancer; Metastatic Esophageal Cancer; Metastatic Gastric Cancer; Cetuximab; Metastatic Esophageal and Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Other): Patients received cetuximab at an initial dose of 400 mg/m2 administered IV over 120 min, followed by weekly infusions at 250 mg/m2 administered IV over 60 min. Once cycle was 4 weeks of therapy. Patients received treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab
  Other Names: erbitux

SUMMARY:
Purpose: There remains a great need for novel therapeutic agents and treatment strategies for advanced esophagogastric cancer. Preclinical and clinical studies have demonstrated increased EGFR expression in a significant proportion of both esophageal and gastric carcinomas. Inactivation of EGFR through use of a monoclonal antibody in preclinical models has resulted in inhibition of tumor growth. Agents designed to block the EGFR pathway have demonstrated disease control among previously treated patients with metastatic esophageal and gastric cancer. The proposed mechanism of action for cetuximab is its ability to effectively disrupt EGFR-mediated signal transduction pathways that ultimately leads to halting cell cycle progression, induces apoptosis, and also inhibits processes important for tumor growth, such as cell invasion and angiogenesis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary - To assess the response rate of single-agent cetuximab in patients with advanced esophageal or gastric cancer who have failed 1-2 prior chemotherapy regimens given in the metastatic setting.

Secondary

* To evaluate the duration of response, progression-free survival and overall survival.
* To assess the safety of cetuximab.

Exploratory

- To assess whether levels of EGFR expression and/or EGFR mutation status correlates with response and toxicity of cetuximab.

STATISTICAL DESIGN:

This study used a two-stage design to evaluate efficacy of cetuximab based on overall response (OR) defined as complete response (CR) or partial response (PR). The null and alternative OR rate were 5% and 15%. If one or more patients enrolled in the stage one cohort (n=20 patients) achieved PR or better than accrual would proceed to stage two (n=16 patients). There was 36% probability of stopping the trial at stage one if the true OR rate was 5%. The probability that the regimen would be considered promising if the true OR rate was 5% was 10% and 80% if the true OR rate was 15%.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable or metastatic stage IV esophageal or gastric adenocarcinoma. Tumors with squamous cell differentiation, including those with a mixture of squamous and adenomatous differentiation, are excluded.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, greater than or equal to 1 cm (longest diameter) by spiral computed tomography (CT) scan or greater than or equal to 2 cm by other radiographic technique. Disease in an irradiated field as only site of measurable disease is acceptable if there has been a clear progression of the lesion.
* Patients must have at least one paraffin block or twenty unstained slides available for analysis of epidermal growth factor receptor (EGFR) status.
* Treatment with 1-2 prior chemotherapy regimens given in the metastatic setting for unresectable or metastatic esophageal or gastric carcinoma.
* ECOG performance status 0-2.
* Life expectancy greater or equal to 12 weeks.
* Age 18 years or older.
* Ability to sign an informed consent document.
* Neutrophils greater than or equal to 1,000/mm3.
* Platelets greater than or equal to 75,000/mm3.
* Serum bilirubin less than or equal to 2.0 mg/dl.
* Serum creatinine less than or equal to 1.5 mg/dl.
* Aspartate aminotransferase (AST or SGOT) less than or equal to 2.5 x upper institutional normal limit.

Exclusion Criteria:

* Pregnant or lactating women. Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days of initiation of therapy. Men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while in this study.
* Subjects should have no other active malignancy other than non-melanoma skin cancer or in-situ cervical carcinoma. A resected cancer (other than in-situ carcinoma) must have demonstrated no evidence of recurrence for at least 3 years.
* Subjects should not have a significant history of cardiac disease, i.e., uncontrolled hypertension; unstable angina; congestive heart failure; myocardial infarction less than 6 months prior to registration; or serious uncontrolled cardiac arrhythmia.
* Subjects must not have received prior cetuximab or other therapy that specifically and directly targets the EGFR pathway. Prior therapy with bevacizumab is permissible.
* Subjects must not have experienced prior severe infusion reaction to a monoclonal antibody.
* Subjects must not have received any chemotherapy regimen or radiation therapy within 28 days prior to study entry.
* Patients must have completed any major surgery 4 weeks or any minor surgery 2 weeks prior to the first infusion of cetuximab. Patients must have fully recovered from the procedure.
* No concurrent use of chemotherapy, radiation, or other investigational agents is allowed while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A. Chan, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - North Shore Medical Center Cancer Center, Peabody, Massachusetts

REFERENCES:
- [Result] Chan JA, Blaszkowsky LS, Enzinger PC, Ryan DP, Abrams TA, Zhu AX, Temel JS, Schrag D, Bhargava P, Meyerhardt JA, Wolpin BM, Fidias P, Zheng H, Florio S, Regan E, Fuchs CS. A multicenter phase II trial of single-agent cetuximab in advanced esophageal and gastric adenocarcinoma. Ann Oncol. 2011 Jun;22(6):1367-1373. doi: 10.1093/annonc/mdq604. Epub 2011 Jan 7. PMID 21217058

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from September 2005 through November 2008.
Period: Overall Study
Arm/Group | Cetuximab
Started | 43
Eligible | 37
Treated | 35
Completed | 0 (Since treatment duration was not fixed, patients were not considered to have completed treatment.)
Not Completed | 43
Not completed — Progressive Disease | 29
Not completed — Death | 1
Not completed — Clinical Deterioration | 4
Not completed — Withdrawal by Subject | 3
Not completed — Ineligible | 6

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of eligible and treated patients.
Arm/Group | Cetuximab
Number analyzed (Participants) | 35
Age, Customized [Median (Full Range); unit: years] | 61 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 35
Primary Tumor [Number; unit: participants]
  Esophagael | 12
  GE Junction | 8
  Gastric | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response (OR) rate was defined as achieving partial response (PR) or complete response (CR) based on RECIST 1.0 criteria on treatment. Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment; Treatment continued until disease progression or unacceptable toxicity. Treatment duration was a median of 6 weeks (range 1-23 weeks).
Population: Responses were determined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Measure: Number (90% Confidence Interval); unit: proportion of paticipants
Arm/Group | Cetuximab
Number analyzed (Participants) | 35
proportion of paticipants | 0.029 [0.0014 to 0.128]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 5/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=35)
Hemoglobin (Blood and lymphatic system disorders) | 1
Lymphocytes (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 2
Headache (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Acneiform Rash (Skin and subcutaneous tissue disorders) | 1
Pruritis/itching (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=35)
Hemoglobin (Blood and lymphatic system disorders) | 16
Leukocytes (Blood and lymphatic system disorders) | 4
Lymphocytes (Blood and lymphatic system disorders) | 7
Platelets (Blood and lymphatic system disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 14
Hyperglycemia (Metabolism and nutrition disorders) | 8
Aspartate aminotransferase (Metabolism and nutrition disorders) | 5
Alanine aminotransferase (Metabolism and nutrition disorders) | 4
Alkaline phosphatase (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Bilirubin (Renal and urinary disorders) | 1
Abdominal pain (General disorders) | 6
Chest pain (General disorders) | 2
Hypersensitivity reaction (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Anorexia (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dehydration (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 20
Fever (General disorders) | 6
Headache (General disorders) | 4
Mucositis (Gastrointestinal disorders) | 4
Nail changes (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 12
Sensory neuropathy (Nervous system disorders) | 2
Acneiform rash (Skin and subcutaneous tissue disorders) | 26
Vomiting (Gastrointestinal disorders) | 8
Weight loss (General disorders) | 4
Rigors/chills (General disorders) | 2
Pruritis/itching (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No